CLINICAL TRIAL: NCT06244966
Title: Verifying Remote Low Volume Blood Tests for Genito-urinary Infections Including Syphilis and Bloodborne Viruses
Brief Title: GUM Remote Testing v4.0
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Royal Devon and Exeter NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2312510
Record Dates: First submitted 2024-01-16; First posted 2024-02-06 (Actual); Last update posted 2024-04-10 (Actual); Status verified 2024-04

CONDITIONS: HIV Infections; Syphilis Infection; Hepatitis B and Hepatitis C
MeSH Terms: conditions — HIV Infections; Hepatitis B; Hepatitis C

STUDY DESIGN:
Intervention Model Description: Comparative study of two collection methods for blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Any client attending clinic for venous blood sampling (Experimental): Any client attending clinic for venous blood sampling for sexually transmitted disease diagnostics will also collect capillary blood using a finger prick
  Interventions: Diagnostic Test: HIV diagnostic testing

INTERVENTIONS:
Diagnostic Test: HIV diagnostic testing — Finger-prick capillary blood will be tested alongside venous blood
  Other Names: Syphilis diagnostic testing; Hepatitis diagnostic testing

SUMMARY:
Capillary blood sample results are compared to venous blood results

DETAILED DESCRIPTION:
Capillary blood samples can be taken by patients from their own finger without requiring a healthcare professional to take a blood sample. Samples taken this way can be posted from home. This crucially avoids visits to the clinic or hospital to have blood samples taken. It would reduce the burden on healthcare professionals and is often preferred by patients. It is important to demonstrate that the results of an analysis performed on capillary blood samples are equivalent to the analysis of a standard venous sample.

This study aims to collect, in parallel to a standard venous blood sample, a capillary blood sample taken by the participant which is then added to specially designed filter paper (dried plasma spot sample) or other collection devices. Parallel analysis of paired samples will then allow the investigators to assess if results measured in samples taken using the two methods are similar.

The investigators will recruit 40 participants for each collection device to this study. It is important to obtain a range of positive and negative results from the study participants, and from stored samples and quality control material.

ELIGIBILITY:
Inclusion Criteria:

* Adults
* Able and willing to provide informed consent.
* Already having a venous blood sample for clinical care

Exclusion Criteria:

* Failure to consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-05 (Estimated); Primary Completion 2025-05 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
Comparative capillary and venous samples screening testing | 1 year
  To have sufficient parallel samples (capillary and venous) collected to demonstrate equivalence of the results of HIV, HBV, HCV and syphilis testing using the Roche Cobas e601 platform

SECONDARY OUTCOMES:
Comparative capillary and venous samples confirmatory testing | 1 year
  To have sufficient parallel samples (capillary and venous) collected to demonstrate equivalence of the results of HIV, HBV, HCV and syphilis testing using other platforms and for viral load

CONTACTS AND LOCATIONS:
Locations (1):
- Royal Devon University Hospital NHS Foundation Trust, Exeter, Devon, United Kingdom

IPD SHARING:
Plan to Share IPD: No
No data will be shared